CLINICAL TRIAL: NCT07140458
Title: Comparative Effect of Box Breathing And Buteyko Breathing on Pulmonary Functions in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0325 Ezaz
Record Dates: First submitted 2025-07-14; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Asthma (Diagnosis); Breathing Exercises
Keywords: Asthma; Breathing Exercise; Buteyko Breathing; Box Breathing; Pulmonary Function tests
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko Breathing (Experimental): Using Buteyko Breathing as primary intervention in addition to standard Asthma therapy.
  Interventions: Other: Buteyko Breathing
- Box Breathing Technique (Experimental): Using Buteyko Breathing as primary intervention in addition to standard Asthma therapy.
  Interventions: Other: Box breathing

INTERVENTIONS:
Other: Buteyko Breathing — Buteyko Breathing is a technique focusing on controlled, reduced breathing to improve oxygen uptake and reduce hyperventilation-related symptoms using Air hunger.
  Procedure:-
  After gaining proper relaxation:
  1. Exhale slowly, and then hold that breath.
  2. Use the index finger and thumb to plug the nose.
  3. Hold that breath until there is an urge to breathe, and then inhale.
  4. Breathe normally for at least 10 seconds.
  5. Repeat several times.
  Arms: Buteyko Breathing
Other: Box breathing — Box Breathing (4-4-4-4 Technique) - Box Breathing exercises boosts lung function by optimizing oxygen flow and activating relaxation responses.Each exercise Sessions included 20 cycles of Box Breathing.
  The procedure of the box breathing cycle includes:
  1. inhale for 4 seconds
  2. Hold the breath for 4 seconds
  3. Exhale for 4 seconds
  4. Hold the breath for 4 seconds, and repeat.
  Arms: Box Breathing Technique

SUMMARY:
The aim of this study was to evaluate the Effectiveness of Box Breathing Technique and Buteyko breathing techniques in patients with Asthma, using both Clinical Pulmonary tests as well as Patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with bronchial asthma for more than one year
* Subjects who are on regular treatment (both inhalers and medication).
* Subjects who are conscious and cooperative.

Exclusion Criteria:

* Subject with recent abdominal, thoracic surgery.
* Subject with any Disability; Physical or Mental.
* Subjects who have other chronic respiratory diseases, new or current smoker, and had respiratory tract infection.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Lung Function tests (FVC) | through study completion, approximately 8 weeks
  Changes from Baseline, Lung function tests measure how well the lungs take in, hold, and move air, as well as how efficiently they transfer oxygen into the blood. These tests help diagnose and monitor respiratory diseases like asthma, COPD, pulmonary fibrosis, and restrictive lung diseases. Tets measures are compared against Normal value i.e: FVC ≥80%.
Lung Function Test (FEV¹) | through study completion, approximately 8 weeks
  Changes from Baseline, Lung function tests measure how well the lungs take in, hold, and move air, as well as how efficiently they transfer oxygen into the blood. These tests help diagnose and monitor respiratory diseases like asthma, COPD, pulmonary fibrosis, and restrictive lung diseases. Test measures are compared against Normal value i.e: FEV¹ ≥80%.
Lung Function test (FEV₁/FVC ratio) | through study completion, approximately 8 weeks
  Changes from Baseline, Lung function tests measure how well the lungs take in, hold, and move air, as well as how efficiently they transfer oxygen into the blood. These tests help diagnose and monitor respiratory diseases like asthma, COPD, pulmonary fibrosis, and restrictive lung diseases. Test measures are compared against Normal value i.e: FEV₁/FVC ≥0.7.

SECONDARY OUTCOMES:
Modified Borg Dyspnea Scale | through study completion, approximately 8 weeks
  The Modified Borg Dyspnea Scale (MBS) is a subjective tool used to measure a patient's perceived breathlessness (dyspnea) during physical activity or at rest.
  Scoring System:
  -Scale Range: 0 to 10(with verbal descriptors for each level). Higher values signify worse condition (Maximal effort).
Mcgill quality of life questionnaire | through study completion, approximately 8 weeks
  The MQOL is a validated tool designed to assess the quality of life (QoL) in patients with life-threatening or chronic illnesses. It focuses on *physical, psychological, existential, and social well-being*.
  Response Scale: Most items use a 0-10 numerical rating scale (higher = better QoL).
  * 0 = Worst possible experience
  * 10= Best possible experience Overall Higher scores indicate better quality of life. Whereas Lower scores suggest significant distress in a domain (e.g., pain, existential crisis).

CONTACTS AND LOCATIONS:
Overall Officials: Qurat ul Ain, Masters, Principal Investigator — Riphah International University
Locations (1):
- Islam center and Teaching Hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Satria O, Apriani F, Damayanti S, Muharamah D. Pengaruh Teknik Pernapasan Buteyko Terhadap Penurunan Kekambuhan Asma Pada Pasien Asma Bronkhial. Journal Of Health And Physical. 2025;1(1):1-7.
- [Background] Abd Allah Abd El Hafeez N, Khalil Hafez M, Mohamed ahmed Z, Metwally El-Sayed M, Abdelwahab Khedr M, Fathy ahmed dawood R. Evaluating the Effect of Buteyko Breathing Technique in Enhancing Asthma Control and Life Quality Among Asthma Patients: A Nursing-Led QuasiExperimental Study. Egyptian Journal of Health Care. 2025;16(1):831-52.
- [Background] Celik H, Yuruk E. The effect of the Buteyko breathing technique on asthma control and quality of life in children with asthma aged 7-12 years: a randomized controlled study. PeerJ. 2025 Jun 3;13:e19467. doi: 10.7717/peerj.19467. eCollection 2025. PMID 40487067
- [Background] Mahmoud Abo El-Fadl N, Mohammed Mahmoud D. Buteyko Breathing Technique versus Pranayama Technique on Asthma Control among Asthmatic Patients. Journal of Nursing Science Benha University. 2024;5(2):728-54
- [Background] Mokkink L, Prinsen C, Patrick D, Alonso J, Bouter L, De Vet H, et al. COSMIN methodology for systematic reviews of Patient-Reported Outcome Measures (PROMs)-User manual (version 1.0). Retrieved from. 2018
- [Background] Crisafulli E, Clini EM. Measures of dyspnea in pulmonary rehabilitation. Multidiscip Respir Med. 2010 Jun 30;5(3):202-10. doi: 10.1186/2049-6958-5-3-202. PMID 22958431
- [Background] Santoso FM, Harmayetty H, Bakar A, editors. PERBANDINGAN LATIHAN NAPAS BUTEYKO DAN UPPER BODY EXERCISE TERHADAP ARUS PUNCAK EKSPIRASI PADA PASIEN DENGAN ASMA BRONKIAL2014.
- [Background] Udayani W, Amin MF, Makhfudli M. The Effect of Combination of Buteyko Breathing Technique and Walking Exercise on Forced Peak Expiratory Flow In Adult Asthmatic Patients. Jurnal Keperawatan Padjadjaran. 2019
- [Background] Vagedes J, Helmert E, Kuderer S, Vagedes K, Wildhaber J, Andrasik F. The Buteyko breathing technique in children with asthma: a randomized controlled pilot study. Complement Ther Med. 2021 Jan;56:102582. doi: 10.1016/j.ctim.2020.102582. Epub 2020 Oct 23. PMID 33197659
- [Background] Ahmed A, Gayatri Devi R, Jothi Priya A. Effect of Box Breathing Technique on Lung Function Test. 2021.
- [Background] Mohamed NK, Sayed EH, Abd-Elhamed AG. Comparison between The Effect of Buteyko and Pranayama Breathing Techniques on Children with Asthma. Assiut Scientific Nursing Journal. 2022;10(29):139-51.
- [Background] Yosifine Y, Margaretha M, Fatik R, Saputra R, Naning D, Meiliana R, et al. Intervensi teknik pernafasan Buteyko terhadap penurunan respirasi rate dan saturasi oksigen pada pasien asma bronchial: Intervention of Buteyko breathing technique on reduction of respiratory rate and oxygen saturation in bronchial asthma patients. Open Access Jakarta Journal of Health Sciences. 2022;1(9):318-22
- [Background] Azab A, Moawd S, AbdulRahman R. Effect of buteyko breathing exercises versus yoga training on pulmonary functions and functional capacity in children with bronchial asthma: a randomized controlled trial. International Journal of Therapies and Rehabilitation Research. 2017;6(1):148.
- [Background] David J, Patil H. Immediate effect of Buteyko breathing technique versus stacked breathing technique in asthma patients. International journal of health science and research. 2022;12(6):158
- [Background] Sankar J, Das RR. Asthma - A Disease of How We Breathe: Role of Breathing Exercises and Pranayam. Indian J Pediatr. 2018 Oct;85(10):905-910. doi: 10.1007/s12098-017-2519-6. Epub 2017 Dec 16. PMID 29247426
- [Background] AbdElmawla Elsaid RA, Zahran WE-k, Elsaid Hafez DM. Comparison of the Effects of Buteyko and Diaphragmatic Breathing Technique on Improving Pulmonary Functions and Asthma Control among Patients with Bro. Egyptian Journal of Nursing and Health Sciences. 2023;4(3):57-75.
- [Background] Hasoon ZK, Abdulwahhab MM. Effectiveness of Buteyko Technique, Pursed-Lip Breathing, and Inhaler Technique Program on Asthma Control for Patients with Asthma. Bahrain Medical Bulletin. 2024;46(
- [Background] Kwa E-K, Cheong S-K, Ong L-K, Lee P-F. Comparing Guided and Non-guided Deep Breathing Impact on Disability Well-Being: A Systematic Review. Journal of Medical and Biological Engineering. 2024;44(5):635-54.
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Kendrick KR, Baxi SC, Smith RM. Usefulness of the modified 0-10 Borg scale in assessing the degree of dyspnea in patients with COPD and asthma. J Emerg Nurs. 2000 Jun;26(3):216-22. doi: 10.1016/s0099-1767(00)90093-x. PMID 10839848
- [Background] Kharaba Z, Feghali E, El Husseini F, Sacre H, Abou Selwan C, Saadeh S, Hallit S, Jirjees F, AlObaidi H, Salameh P, Malaeb D. An Assessment of Quality of Life in Patients With Asthma Through Physical, Emotional, Social, and Occupational Aspects. A Cross-Sectional Study. Front Public Health. 2022 Sep 1;10:883784. doi: 10.3389/fpubh.2022.883784. eCollection 2022. PMID 36117601
- [Background] Lisspers K, Stallberg B, Hasselgren M, Johansson G, Svardsudd K. Quality of life and measures of asthma control in primary health care. J Asthma. 2007 Nov;44(9):747-51. doi: 10.1080/02770900701645298. PMID 17994405
- [Background] Feeny DH, Eckstrom E, Whitlock EP, Perdue LA. A Primer for Systematic Reviewers on the Measurement of Functional Status and Health-Related Quality of Life in Older Adults [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2013 Sep. Report No.: 13-EHC128-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK169159/ PMID 24199257
- [Background] Expert Panel Working Group of the National Heart, Lung, and Blood Institute (NHLBI) administered and coordinated National Asthma Education and Prevention Program Coordinating Committee (NAEPPCC); Cloutier MM, Baptist AP, Blake KV, Brooks EG, Bryant-Stephens T, DiMango E, Dixon AE, Elward KS, Hartert T, Krishnan JA, Lemanske RF Jr, Ouellette DR, Pace WD, Schatz M, Skolnik NS, Stout JW, Teach SJ, Umscheid CA, Walsh CG. 2020 Focused Updates to the Asthma Management Guidelines: A Report from the National Asthma Education and Prevention Program Coordinating Committee Expert Panel Working Group. J Allergy Clin Immunol. 2020 Dec;146(6):1217-1270. doi: 10.1016/j.jaci.2020.10.003. PMID 33280709
- [Background] Reddel HK, Bacharier LB, Bateman ED, Brightling CE, Brusselle GG, Buhl R, Cruz AA, Duijts L, Drazen JM, FitzGerald JM, Fleming LJ, Inoue H, Ko FW, Krishnan JA, Levy ML, Lin J, Mortimer K, Pitrez PM, Sheikh A, Yorgancioglu AA, Boulet LP. Global Initiative for Asthma Strategy 2021: executive summary and rationale for key changes. Eur Respir J. 2021 Dec 31;59(1):2102730. doi: 10.1183/13993003.02730-2021. Print 2022 Jan. PMID 34667060
- [Background] Jassam AK, Hassan HS. The Effectiveness of a Self-Care Instructional Program on the HealthRelated Quality of Life for Patients with Permanent Pacemaker in Baghdad Teaching Hospitals. Journal of Cardiovascular Disease Research. 2021;12(3):1056-74.
- [Background] Evaristo KB, Mendes FAR, Saccomani MG, Cukier A, Carvalho-Pinto RM, Rodrigues MR, Santaella DF, Saraiva-Romanholo BM, Martins MA, Carvalho CRF. Effects of Aerobic Training Versus Breathing Exercises on Asthma Control: A Randomized Trial. J Allergy Clin Immunol Pract. 2020 Oct;8(9):2989-2996.e4. doi: 10.1016/j.jaip.2020.06.042. Epub 2020 Aug 6. PMID 32773365
- [Background] Manikonda P, Stoerk S, Toegel S, Schardt F, Angermann C, Gruenberger I, et al. P-232: Influence of non-pharmacological treatment (contemplative meditation and breathing technique) on stress induced hypertension-a randomized controlled study. American Journal of Hypertension. 2005;18(S4):89A-90A
- [Background] Zaccaro A, Piarulli A, Laurino M, Garbella E, Menicucci D, Neri B, Gemignani A. How Breath-Control Can Change Your Life: A Systematic Review on Psycho-Physiological Correlates of Slow Breathing. Front Hum Neurosci. 2018 Sep 7;12:353. doi: 10.3389/fnhum.2018.00353. eCollection 2018. PMID 30245619
- [Background] Arora RD, Subramanian VH. To study the effect of Buteyko breathing technique in patients with obstructive airway disease. International Journal of Health Sciences and Research. 2019;9(3):50-64.
- [Background] Hassan EEM, Abusaad FE, Mohammed BA. Effect of the Buteyko breathing technique on asthma severity control among school age children. The Egyptian Journal of Bronchology. 2022;16(1):45.
- [Background] Villareal GMC, Villazor BPU, Villegas AM, Visaya P, Vista ME, Tan CB, et al. Effect of Buteyko method on asthma control and quality of life of Filipino adults with bronchial asthma. The Journal of Macro Trends in Health and Medicine. 2014;2(1):44-60.
- [Background] Santino TA, Chaves GS, Freitas DA, Fregonezi GA, Mendonca KM. Breathing exercises for adults with asthma. Cochrane Database Syst Rev. 2020 Mar 25;3(3):CD001277. doi: 10.1002/14651858.CD001277.pub4. PMID 32212422
- [Background] Sarvesh S, Koushik Muthu Raja M, Rajanandh MG, Seenivasan P. Prevalence and pattern of usage of complementary and alternative medicine among south Indian asthma patients in a tertiary care hospital. Complement Ther Clin Pract. 2018 Feb;30:103-108. doi: 10.1016/j.ctcp.2017.12.016. Epub 2017 Dec 21. PMID 29389468
- [Background] Bhatia R, Abu-Hasan M, Weinberger M. Exercise-Induced Dyspnea in Children and Adolescents: Differential Diagnosis. Pediatr Ann. 2019 Mar 1;48(3):e121-e127. doi: 10.3928/19382359-20190219-02. PMID 30874820
- [Background] Aalbers R, Vogelmeier C, Kuna P. Achieving asthma control with ICS/LABA: A review of strategies for asthma management and prevention. Respir Med. 2016 Feb;111:1-7. doi: 10.1016/j.rmed.2015.11.002. Epub 2015 Nov 6. PMID 26614594
- [Background] Shafiek H. Inhaled Corticosteroids: Benefits and Risks. Updates on Corticosteroids: IntechOpen; 2023.
- [Background] Cates CJ, Jaeschke R, Schmidt S, Ferrer M. Regular treatment with salmeterol and inhaled steroids for chronic asthma: serious adverse events. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD006922. doi: 10.1002/14651858.CD006922.pub3. PMID 23543548
- [Background] Amirav I, Garcia G, Le BK, Barria P, Levy G, Aggarwal B, Fahrbach K, Martin A, Phansalkar A, Sriprasart T. SABAs as Reliever Medications in Asthma Management: Evidence-Based Science. Adv Ther. 2023 Jul;40(7):2927-2943. doi: 10.1007/s12325-023-02543-9. Epub 2023 Jun 7. PMID 37280414
- [Background] Colledge NR, Walker BR, Ralston S, Davidson LSP. Davidson's principles and practice of medicine. (No Title). 2014.
- [Background] Hassan ZM, Riad NM, Ahmed FH. Effect of Buteyko breathing technique on patients with bronchial asthma. Egyptian Journal of Chest Diseases and Tuberculosis. 2012;61(4):235-41.
- See also: Global Strategy for Asthma Management and Prevention. [Online Web Data]. 2023 — https://ginasthma.org/